CLINICAL TRIAL: NCT00545727
Title: Blood Glucose Response to Meals of Varying Glycemic Index in Youth With Type 1 & 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 06-CH-N182
Record Dates: First submitted 2007-10-16; First posted 2007-10-17 (Estimated); Last update posted 2007-10-17 (Estimated); Status verified 2007-09

CONDITIONS: Type 1 Diabetes; Type 2 Diabetes; Impaired Glucose Metabolism
Keywords: Diabetes; Children; Adolescents; Diet; Glycemic index
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HGI (Other): High/standard glycemic index diet
  Interventions: Other: Standard diet
- LGI (Experimental): Low glycemic index diet
  Interventions: Behavioral: Diet

INTERVENTIONS:
Behavioral: Diet — Whole-foods, low glycemic index diet
  Arms: LGI
Other: Standard diet — Standard diet meeting American Diabetes Association guidelines
  Arms: HGI

SUMMARY:
Research to date suggests that the selection of lower glycemic index foods, that is, foods provoking a slower, more sustained blood sugar response, may result in improved glycemic control in youth with diabetes. However, there is currently insufficient data to support practice recommendations. The purpose of this pilot study is to test the blood glucose response to low and high glycemic index meals in youth with diabetes using continuous blood glucose monitoring, and to determine whether the effect of glycemic index differs by regimen or diagnosis. In this pilot study up to 42 youth with type 1 diabetes or impaired glucose metabolism (elevated fasting glucose, insulin resistance, or type 2 diabetes) will participate in 5 days of continuous blood glucose monitoring during which they will receive both low and high glycemic index meals. Children will be provided with 1 full day of low glycemic index meals and 1 full day of high glycemic index meals in a supervised setting in randomized order. Each of these test days will be preceded by a standard evening meal and snack. Continuous blood glucose monitoring will also be conducted during regular food intake ad libidum away from the clinic, as well as during one day of instructed low glycemic meals at home. All food intake, insulin, and blood glucose self-monitoring will be recorded. While in the clinic, measures of satiety and acceptability of the food will also be obtained. Data analysis will include indices of blood glucose levels and variability.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with type 1 diabetes for a minimum of 1 year with insulin dose greater than or equal to 0.5 u/kg/day, or diagnosed with elevated fasting glucose, insulin resistance, or type 2 diabetes
* age 7 to 16

Exclusion Criteria:

* dietary restrictions that would preclude eating the study diet
* comorbid chronic illness requiring daily medical management
* comorbid major psychiatric diagnosis
* non-English speaking/writing

Ages: 7 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2006-07; Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Blood glucose level

CONTACTS AND LOCATIONS:
Overall Officials: Tonja R. Nansel, PhD, Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)